CLINICAL TRIAL: NCT00000235
Title: Alternate Day Buprenorphine Administration, Phase XII
Brief Title: Alternate Day Buprenorphine Administration, Phase XII - 17
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Vermont (Other)
Model: Crossover | Purpose: Treatment
Other Study IDs: NIDA-06969-17; R01-06969-17
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 2002-12

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to determine if six times daily buprenorphine dose is effective in achieving 120 hour buprenorphine dosing.

ELIGIBILITY:
Please contact site for information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0

PRIMARY OUTCOMES:
Drug use
Opioid withdrawal
Opioid agonist effects
Dose choice

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States